CLINICAL TRIAL: NCT05759624
Title: Evaluation of Vesiculogenesis in Children With GH Deficiency Undergoing Hormone Replacement Therapy
Brief Title: Vesiculogenesis in Children With GH Deficiency (VESCIGHTP)
Acronym: VESCIGHTP
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C211
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: GH Deficiency
Keywords: Growth; GH deficiency; Children; Short stature; Extracellular vescicles
MeSH Terms: conditions — Dwarfism, Pituitary; Dwarfism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/plasma samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hormone replacement therapy with rhGH
  Interventions: Drug: rhGH

INTERVENTIONS:
Drug: rhGH — Hormone replacement therapy with rhGH at a dose of 0.025-0.035 mg/kg of body weight per day (or 0.7-1.0 mg/m2 of body surface area per day).

SUMMARY:
The primary objective of the study is to evaluate the size and derivational profile of the extracellular vescicles (EV) generated in children with GH deficiency, undergoing hormone replacement therapy with rhGH. Secondary objectives is to correlate vesiculogenesis with auxometric and biochemical parameters used in clinical-endocrine practice in the evaluation of short stature.

The results of the study will provide useful information to more rationally set up the clinical and biochemical follow-up of hormone replacement therapy with rhGH, as well as to understand the molecular and cellular mechanisms underlying the multi-systemic action of GH, the most important anabolic hormone of the human organism.

DETAILED DESCRIPTION:
Methods:

At the Regional Reference Center for Growth Disorders, Istituto Auxologico Italiano, IRCCS, Milan, 10 children of both sexes affected by isolated GH deficiency will be recruited according to the criteria set out in AIFA note 39 for this pathology (short stature: ≤ - 3 SD or ≤ -2 SD and growth velocity/year ≤ -1.0 SD for age and sex evaluated at least 6 months apart and peak GH at two different stimulating pharmacological tests < 8 ng/ml). The exclusion criterion from the present study (and from treatment with rhGH) will be the presence of organic pathologies at the hypothalamic-pituitary level (assessed by brain MRI).

In basal conditions (pre-treatment), we will proceed with the collection of clinical and anthropometric/auxometric data, including the evaluation of body composition with bioimpedance analysis. The same work-up will be repeated at the subsequent 6-month follow-up (see below).

Each subject will undergo hormone replacement therapy with rhGH at a dose of 0.025-0.035 mg/kg of body weight per day (or 0.7-1.0 mg/m2 of body surface area per day).

In conditions of fasting (at least 12 hours), blood samples will be taken at T0 (i.e., before the start of hormone replacement therapy with rhGH) and at T6 (i.e., after 6 months of rhGH, approximately 10-12 hours after administration of the previous day's dose).

In the samples taken at T0 and T6, the dimensional and derivational profiles of the EVs will be determined. Markers for the following cell subtypes will be identified: endothelium (activated and not), monocytes, neutrophils, platelets, muscle, bone, and adipose tissue.

In basal conditions (T0) and at T6 the patients will be sampled for the determination of the following parameters: complete blood count + formula, blood glucose, insulin, glycated Hb, triglycerides, total cholesterol, LDL, HDL, hsPCR, IGF-1, osteocalcin, ICTP, and PIIIINP.

Quantitative data will be expressed as mean ± SD or as median with interquartile range (Q1-Q3), as appropriate. Categorical data will be presented as frequencies and percentages, while continuous variables will be tested for normality and linearity. If appropriate, a log transformation of the data will be performed. The paired Student's t-test (or other non-parametric test) will be used to compare demographic, clinical, and biochemical characteristics among the same subjects at T0 vs. T6. EVs will be subdivided according to their size (exosomes, microvesicles, and total EVs) and their cellular origin identified by specific markers (e.g., CD14+, CD61+, CD62E+, CD105+, SCGA+, FABP+, etc). Multiple linear regression analysis will be applied to evaluate the association between EVs (as Δ% between T0 and T6 for the dimensional and also derivational profile), circulating IGF-1 levels (as Δ% between T0 and T6), and the rate of growth (T0 to T6). In addition, a paired Student t-test will be used to assess the rhGH-induced change in EV (T0 vs. T6). The test will be applied for all EV populations studied with the size profile and for all vesicular markers studied with the derivational profile. Alternatively, a non-parametric test will be applied. A p-value < 0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* short stature: ≤ - 3 SD or ≤ -2 SD
* growth velocity/year ≤ -1.0 SD for age and sex evaluated at least 6 months apart - peak GH at two different stimulus pharmacological tests < 8 ng/ml

Exclusion Criteria:

- presence of organic pathologies at the hypothalamic-pituitary level (assessed by performing brain MRI).

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 10 children of both sexes affected by isolated GH deficiency will be recruited according to the criteria set out in AIFA note 39 for this pathology (short stature: ≤ - 3 SD or ≤ -2 SD and growth velocity/year ≤ -1.0 SD for age and sex evaluated at least 6 months apart and peak GH at two different stimulus pharmacological tests < 8 ng/ml).
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Size of extracellular vesicles | Baseline and after 6 months
  Change in size of extracellular vesicles after rhGH treatment
Derivational profile of extracellular vesicles | Baseline and after 6 months
  Change in derivational profile of extracellular vesicles after rhGH treatment

SECONDARY OUTCOMES:
Auxometric parameters - height | Baseline and after 6 months
  Change in height after rhGH treatment
Auxometric parameters - weight | Baseline and after 6 months
  Change in weight after rhGH treatment
Biochemical parameters - glycemia | Baseline and after 6 months
  Change in glycemia after rhGH treatment
Biochemical parameters - Insulin-like growth factor I (IGF-I) | Baseline and after 6 months
  Change in IGF-I after rhGH treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy